CLINICAL TRIAL: NCT04519346
Title: Comparison of Intradermal Mesotherapy With Systemic Therapy in the Treatment of Migraine Headache: A Prospective Randomized Study
Brief Title: Mesotherapy Versus Systemic Therapyin Treatment of Migraine Headache
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ataturk University (Other)
Responsible Party: Principal Investigator, Abdullah Osman KOCAK, Principal Investigator, Ataturk University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AtaturkU0002
Record Dates: First submitted 2020-08-17; First posted 2020-08-19 (Actual); Last update posted 2020-08-19 (Actual); Status verified 2020-08

CONDITIONS: Migraine Headache
Keywords: Mesotherapy; Migraine
MeSH Terms: conditions — Migraine Disorders | interventions — Injections, Intradermal

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Compare to sistemic treatment and mesotherapy. (Other): This is a prospective parallel randomized controlled trial conducted with patients admitted to our emergency department with migraine pain
  Interventions: Other: intradermal injection

INTERVENTIONS:
Other: intradermal injection — Mesotherapy was performed by an experienced and trained physician using disposable 4 mm and 6 mm long 30 Gauge needles (Meso-relle, Biotekne SRL, Italy)to the pericarotid region, glabella, and the area between the eyes and ears, and to the area of the head where pain occurred (such as frontal, parietal, occipital region) for each patient

SUMMARY:
Introduction:Migraine is a prevalent disabling primary headache disorder which is classified in two major types; migraine without aura and migraine with aura. The aim of this study was to compare the efficiency of mesotherapy with systemic therapy in pain controlin patients with headache related tomigraine without aura.

Methods: We conducted this prospective parallel randomized controlled trial with the patients admitted to the emergency department with headache related to migraine without aura. One group was treated with mesotherapy, and the control group with intravenous dexketoprofen. Changes in pain intensity at 30th minute, 60th minute, 120th minute and 24th hours after treatment using Visual Analogue Scale (VAS), need to use analgesic drug within 24 hours,re-admission with same complaint to emergency department (ED) within 72 hours, and adverse effect rate of the methods were compared between groups.

ELIGIBILITY:
Inclusion Criteria:

* 18 years and older age, and (2)
* Admission to Emergency Department (ED) with headache related to the migraine without aura.

Exclusion Criteria:

* Taking analgesic drugs before admission,
* Having VAS score of lower than 4 on admission,
* Having diabetes mellitus,
* Body mass index>30 kg/m2,
* Pregnancy,
* Lactation,
* Having active bleeding or bleeding disorder,
* Having active or recurrent gastrointestinal hemorrhage or ulcer, or history of these conditions,
* Having a serious or life-threatening condition (stroke, intracranial hemorrhage, heart attack, cardiac tamponade, pneumothorax, hemothorax, flail chest, etc.).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Actual)
Dates: Start 2019-12-01 (Actual); Primary Completion 2020-02-29 (Actual); Study Completion 2020-05-01 (Actual)

PRIMARY OUTCOMES:
change in headache intensity | 0-24 hours
  Visual Analog Score(points between 0-10. the most severe pain 10 points, no pain 0 points) scores at 30th, 60th and 120th minutes, and 24th hours from the baseline VAS score (at the beginning of the treatment).
need to use analgesics within 24 hours after treatment | 0-24 hours
  We defined this as a requirement of any type analgesics for painkilling at any time within 24 hours of treatment, and this was evaluated by patients, subjectively. we will learn by asking by phone.

CONTACTS AND LOCATIONS:
Locations (1):
- Ataturk University, Erzurum, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Akbas I, Kocak MB, Kocak AO, Gur STA, Dogruyol S, Demir M, Cakir Z. Intradermal mesotherapy versus intravenous dexketoprofen for the treatment of migraine headache without aura: a randomized controlled trial. Ann Saudi Med. 2021 May-Jun;41(3):127-134. doi: 10.5144/0256-4947.2021.127. Epub 2021 Jun 1. PMID 34085549